CLINICAL TRIAL: NCT02739555
Title: Non-inferiority Trial of Three Cycles of Zoledronic Acid Versus Percutaneous Thermal Ablation in Osteoid Osteoma
Brief Title: Zoledronic Acid Compared to Percutaneous Treatment in Osteoid Osteoma
Acronym: BISPHOO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study has been conducted until the end of the research; participants are no longer receiving an intervention or being examined; but recruitment isn't completed (15 % enrolled in the stud)
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140909; 2015-001698-41 (EudraCT Number)
Record Dates: First submitted 2016-03-29; First posted 2016-04-15 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Osteoid Osteoma
Keywords: Osteoid osteoma; Bisphophonates
MeSH Terms: conditions — Osteoma, Osteoid | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Percutaneous treatment (Active Comparator): Percutaneous treatment of OO is a thermal tumor destruction by radiofrequency or laser photocoagulation performed under CT control with strict aseptic approach and most often under general anesthesia. The introductive needle is inserted toward the nidus. Then the optic fiber or the radiofrequency probe is inserted in the nidus center and thermal destruction of the tumor is obtained.When the distance between the nidus and a nerve or the skin is less than 10 mm, infusion of normal saline or CO2 is introduced as spacing agent. When the nidus is in the subchondral bone, cold normal saline is introduced in the joint to protect the cartilage. In addition, a thermocouple is placed in the epidural or foraminal space to continuously monitor the temperature. A procedure typically required between 1 and 2 h from the time the patient entered the CT unit.
  Interventions: Device: Thermal destruction with radiofrequency or laser
- 2: Bisphosphonate treatment (Experimental): The treatment consists of 3 infusions of zoledronic acid administered at a monthly interval. Bisphosphonate treatment is considered finished 1 month after the third bisphosphonate infusion (V4 visit). In few cases, the analgesic efficacy provided by 3 bisphosphonate infusions cannot be sufficient: 1 to 3 additional infusions could be proposed to the patient.
  Zoledronic acid is supplied as a 4 mg/100 ml solution for infusion. It will be administered as infusion over 30 minutes under the supervision of a nurse. Adults will receive intravenous infusion of 4 mg of zoledronic acid. Children will receive infusion of 0.025 mg/kg of zoledronic acid.
  The investigators propose abacus corresponding to zoledronic acid volume to infuse during 30 minutes for children.
  Interventions: Drug: Acide Zoledronique

INTERVENTIONS:
Device: Thermal destruction with radiofrequency or laser
  Arms: 1: Percutaneous treatment
Drug: Acide Zoledronique
  Arms: 2: Bisphosphonate treatment

SUMMARY:
Osteoid osteoma (OO) is a benign osteogenic tumor occurring in children and young adults, responsible for intense bone pain, which has a tendency to spontaneously heal with mineralization of the nidus, but extremely slowly. This healing may be accelerated in patients taking NSAIDs regularly during a few years. The long delay for healing and intense pain, explain why patients are quickly directed to surgeons or specialized radiology departments for tumor ablation. But percutaneous treatment or surgical excision destruction can expose the patient to a substantial risk in terms of neurologic or joint damages, depending on the location. Bisphosphonates treatment may be an effective alternative to percutaneous treatment by accelerating the natural history of OO.

DETAILED DESCRIPTION:
Osteoid osteomas (OOs) are small, benign but painful bone tumors, mainly observed in children and young adults. Pain, almost universal, is characteristically greater at night. Pain is well relieved by NSAIDs but resolution is not always complete and pain reappears a few hours after the last dose. Also long-term consumption of NSAID can lead to serious adverse events. Therefore OOs are usually cured shortly after diagnosis, mainly by means of percutaneous treatment (PT) under computed tomography (CT) (radiofrequency coagulation or interstitial laser ablation).

The clinical success rate using these techniques is 96% at 6-month, 94% at 24-month. However, the technique is not distributed everywhere since it is performed by highly specialized interventional radiologists. The PT is performed under general, spinal or regional anesthesia. General anesthesia is used in most cases, especially in children. When the OO is located in close proximity to the skin, cartilage, vessels and nerves, severe complications may occur and additional procedures such as infusion of saline or injection of CO2 at the interface between the OO and the vulnerable structure are done. Also few anatomic locations are not accessible to a PT.

The natural history of OOs remains poorly understood. However investigators in small series of conservatively treated OOs suggested a spontaneous healing of the lesion with mineralization of the nidus and resolution of pain (mean duration of pain in patients with NSAID treatment: 33 months NSAID).

The efficacy of bisphosphonates on pain related to benign (Langherhans cell histiocytosis, fibrous dysplasia, Paget disease) or malignant bone lesions has been widely reported. The investigators observed such efficacy in a small series of 20 patients with percutaneously hard-to-reach or recurrent OO using one to three infusions of zoledronate. The clinical efficacy assessed on pain relief was accompanied by a significantly increased mineralization of the nidus. The investigators postulated that bisphosphonates had accelerated the natural history of OO.

Our hypothesis is that three infusions of zoledronate (4mg) repeated monthly in patients with symptomatic OO is non-inferior to percutaneous treatment on the efficacy, measured by pain relief at Visual Analogical Scale (VAS).

The main objective of this randomized study is to demonstrate that in patients with OO, treatment with three intravenous cycles of 4mg of zoledronic acid administered monthly, is non-inferior to treatment with percutaneous thermal ablation on the efficacy measured by the percentage of pain relief between baseline and end of treatment.

NB: Patients for whom the OO would not be percutaneously accessible (that is to say when the percutaneous treatment or surgical excision destruction expose the patient to a substantial risk in terms of neurologic or joint damages) will be offered to participate in a cohort, only in Lariboisière and Cochin hospital in Paris. In the cohort, the clinical follow-up will be conducted as it is currently proposed in Laribosisière hospital (no act added by the research). Objectives of the register will be explained to the patient. It consists in collecting anonymized medical data after a bisphosphonate treatment to statuate on the efficacy of the bisphosphonates to relieve pain due to osteoid osteoma.

Study design of the randomized study:

* Selection / Inclusion visit: verification of eligibility, randomization and recollection of patient consent.
* Intervention:

  * percutaneous thermal ablation at V1 visit (i.e. maximum one month after the selection / inclusion visit)
  * or three zoledronic acid infusions at V1, V2 (one month after v1) and V3 visits (one month after V2)
* V4 visit at 4 months (end of treatment, evaluation of the main outcome) and V7 visit at 16 months (end of study, evaluation of the secondary outcomes).
* Option: One to 3 additional visits (V4, V5 and V6) for zoledronic acid infusion can be proposed to the patient, depending on the efficacy of the previous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age superior or equal to 10 years
* Patient with a typical osteoid osteoma diagnosed on clinical and radiological criteria (MRI and scanner), validated by a binomial clinician / radiologist.
* OO never treated or in treatment failure, or recurrent OO.
* OO percutaneously accessible
* Pain intensity is superior or equal to 40 mm on a VAS at inclusion visit.
* Written informed consent signed by the patient or his representative (for minors, agreement of the child and signature of the two mandatory parents).
* Patient affiliated to the social security.

Exclusion Criteria:

* Patients with other diseases or receiving treatment that may impact on bone tissue or its metabolism.
* Patients suffering from renal failure (i.e. lower than 60 ml/min according to the Cowcroft equation).
* Patients with severe hepatocellular insufficiency (TP<50%).
* Patients with a history of iritis or uveitis.
* Patient with untreated rickets or osteomalacia.
* Patient with untreated dental infection or planed dental surgery during the study period.
* Patient with untreated infection of the external auditory canal (ex: furuncle, eczema superinfection)
* Patient already treated by bisphosphonates.
* Patients with hypersensitivity to the active substance, to other bisphosphonates or to any of the excipients (List of excipients: mannitol (E421), sodium citrate (E331), water for injections).
* Patient enrolled in another biomedical research protocol and during the whole study
* Pregnant or breastfeeding women, or planning pregnancy during the course of the study
* Women of child bearing potential (women following menarche and until post-menopause) and sexually active, without an effective contraceptive measure during the period of treatment (hormonal contraception or mechanical contraception)*

  * Oral contraceptive methods include:
* combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravagina or transdermal)
* progestogen-only hormonal contraception associated with inhibition of ovulation (oral, intravagina or transdermal).

  * Mechanical methods of contraception include intrauterine device and intrauterine hormone-releasing system.Patient enrolled in another biomedical research protocol and during the whole study

Patients who would not meet the inclusion criteria "OO percutaneously accessible" will be offered to participate in a register, only in Lariboisière hospital. This register will target specifically children aged of at least 12 years old and adults.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Percentage of decrease in bone pain measured on a visual analog scale (VAS) between baseline and the end of treatment larger or equal to 70%. | 4 months
  Percentage of decrease in bone pain measured on a visual analog scale (VAS) between baseline and the end of treatment larger or equal to 70%. End of treatment is set at one month after the third administration of bisphosphonates and three months after the percutaneous thermal destruction (ie 4 months after inclusion visit = V4 visit, for both groups).

SECONDARY OUTCOMES:
Pain | at 1, 2, 3, 7, 10 and 16 months
  arm1 : only at 16 months
  arm 2 : assessed by Visual Analog Scale as an average over the past 48 hours, at V1 (1 month +/- 5 days), V2 (2 months +/- 5 days), V3 (3 months +/- 5 days), V7 visits (16 months +/- 1 month) and, in case of additional infusions, at V5 (7 months +/- 15 days) and V6 (10 months +/- 15 days)
Patient'Global Impression of change (PGIC) | at 2, 3, 7, 10 and 16 months
  arm1 : only at 16 months
  arm 2 : assessed by Visual Analog Scale as an average over the past 48 hours, at V2 (2 months +/- 5 days), V3 (3 months +/- 5 days), V7 visits (16 months +/- 1 month) and, in case of additional infusions, at V5 (7 months +/- 15 days) and V6 (10 months +/- 15 days)
Consumption of analgesic and NSAIDs | at inclusion, 1, 2, 3, 4, 7, 10 and 16 months
  To this end, patient will be asked to note any analgesic and NSAIDs medication in a CRJ during the whole study arm1 : only at inclusion, 1, 4 and16 months
Nidus mineralization on CT scan images | 4 months
Surface of bone marrow edema on MR images | at 4 and 16 months
Incidence of Treatment-Emergent Adverse Events of bisphosphonates and percutaneous treatment. | at inclusion, 1, 2, 3, 4, 7, 10 and 16 months
  Tolerance and adverse events of bisphosphonates and percutaneous treatment. To this end, patient will be asked to note any adverse event in a CRJ during the whole study.
  arm1 : only at inclusion, 1, 4 and16 months

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BOUSSON, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (16):
- France (16):
  - Hopital PELLEGRIN - Service d'imagerie diagnostique et interventionnelle de l'adulte, Bordeaux
  - Hopital PELLEGRIN - Service rhumatologie, Bordeaux
  - Hôpital ROGER SALENGRO - Service d'Orthopédie A, Lille
  - Hôpital ROGER SALENGRO - Radiologie et imagerie musculo-squelettique, Lille
  - Hôpital ROGER SALENGRO - Rhumatologie, Lille
  - Hôpital LAPEYRONIE - Imagerie médicale, Montpellier
  - Hôpital LAPEYRONIE - Service Rhumatologie, Montpellier
  - CHU Nancy - Imagerie Guilloz, Nancy
  - Hôpital LARIBOSISIERE - Service radiologie ostéo-articulaire, Paris
  - Hôpital LARIBOSISIERE - Service rhumatologie, Paris
  - Hôpital COCHIN - Service radiologie B, Paris
  - Hôpital COCHIN - Service rhumatologie B, Paris
  - Hopital SUD - Service Radiologie, Rennes
  - Hôpital SUD - Service rhumatologie, Rennes
  - Hôpital PURPAN - Serice Radiologie, Toulouse
  - Hôpital PURPAN - Serice Rhumatologie, Toulouse

IPD SHARING:
Plan to Share IPD: No